CLINICAL TRIAL: NCT05744024
Title: Non-pharmacological Pain Care Using Virtual Reality Therapy or Music Therapy During Complex Wound Care in Adults
Brief Title: Non-pharmacological Pain Care During Complex Wound Care Procedures
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Marlies P. Schijven, Professor doctor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NL82062.018.22
Record Dates: First submitted 2022-12-12; First posted 2023-02-24 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Wound Surgical; Wounds and Injuries; Virtual Reality; Wound Care; Music Therapy
MeSH Terms: conditions — Surgical Wound; Wounds and Injuries

STUDY DESIGN:
Masking Description: Randomization will not be blinded since both the provider and patient know if the patient will be wearing the VR system or headphone with audio during wound care or not wearing the VR system or headphone with audio.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Virtual Reality Therapy (Intervention group 1) (Experimental): In addition to the standard wound care procedure, the Virtual Reality Therapy group (intervention group 1) will receive the VR system during the wound care. The VR system consists of Virtual Reality glasses, a controller and a headphone. The application SyncVR Relax & Distract will be used, which will contain various videos for the patient those from to relax and be distracted. This group wears the VR system 10 minutes before the start of the wound care, until 1 minute after the wound care has ended.
  Interventions: Device: Virtual Reality system
- Music Therapy (Intervention group 2) (Experimental): In addition to the standard wound care procedure, the Music Therapy group (intervention group 2) will be hearing their preferred audio, chosen by patient to be relaxing and to offer distraction, through headphones during wound care. This group wears the headphone with music 10 minutes before the start of the wound care, until 1 minute after the wound care has ended.
  Interventions: Other: Headphones
- Care as usual (control group/group 3) (No Intervention): The care as usual group (control group) will receive the care as usual. This group receives neither VRT nor MT during wound care.

INTERVENTIONS:
Device: Virtual Reality system — The intervention group 1 will be wearing the 'SyncVR' Virtual Reality system during the wound care moment in addition to the standard procedure. The VR system consists of Virtual Reality glasses, a controller, and a headphone. The SyncVR Relax & Distract Application (SyncVR R&D) will be used.
  Arms: Virtual Reality Therapy (Intervention group 1)
Other: Headphones — Headphones with audio. The patients will be hearing their preferred audio, chosen by patient to relaxing and to offer distraction, through headphones during wound care.
  Arms: Music Therapy (Intervention group 2)

SUMMARY:
The main objective of this study is to evaluate the effect on pain and both Virtual Reality and Music Therapy as add-on therapy during wound car in adults.

DETAILED DESCRIPTION:
After inclusion and completion of the informed consent form, patients are randomly allocated to the intervention group or control group in a 1:1:1 ratio. Randomization will not be blinded since both the provider and patient know if the patient will be wearing the VR system or headphone with audio during wound care or not wearing the VR system or headphone with audio.

Patients are randomly assigned to one of three groups:

Group 1 - Intervention group 1, Virtual Reality Therapy Group 2 - Intervention group 2, Music Therapy Group 3 - Control group, care as usual

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 or older who have wounds receiving wound care
* Individuals who will undergo minimum of 1 to a maximum of 3 sequential complex wound care procedures before discharge
* At least 1 prior painful wound care procedure, where they have indicated a VAS ≥ 4, or patients reporting a VAS ≥ 4 before initiating the wound care procedure.

Exclusion Criteria:

* Individuals not being able to understand Dutch language at primary school level
* Individuals not being able to read or write Dutch
* Individuals diagnosed with dementia and/or cognitive impairment
* Individuals diagnosed with epilepsy
* Individuals diagnosed with migraine
* Individuals with severe dizziness and/or nausea
* Individuals with a known history of claustrophobia
* Individuals who are unable to sign informed consent owing to mental disorder or formally stated to be incompetent to decide
* Individuals who have no feeling in the wound care area
* Individuals with physical (and/or cognitive) disabilities on the face, eye, ear, nose and neck that prevent the use of the VR headgear and/or headphones

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2025-11-17 (Estimated); Study Completion 2025-11-17 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the change in pain score before and after the first wound care, measured with the Visual Analogue Scale (VAS). | Baseline, during the procedure, immediately after procedure
  The VAS is a horizontal scale from 0 to 10, with 0 indicating ''no pain'' and 10 indicating ''worst pain possible''.

SECONDARY OUTCOMES:
Mean VAS change of all wound care procedures included in the study | Baseline, during the procedure, immediately after procedure
  The VAS is a horizontal scale from 0 to 10, with 0 indicating ''no pain'' and 10 indicating ''worst pain possible''.
Change from baseline in level of anxiety at 10 minutes after procedure | Baseline, 10 minutes after procedure
  Level of anxiety, as measured by a Dutch translated and validated modification of the Spielberger State-Trait Inventory-6 (STAI-6) questionnaire 10 minutes before and 10 minutes after each three wound care moments.
Patient satisfaction | Through study completion, an average of 1 week
  Patient satisfaction, as measured by a self-developed Dutch provider satisfaction questionnaire, focuses on satisfaction about the intervention with the VR system or headphone with audio. The questionnaires included a Visual Analogue Scale (VAS). The VAS is a horizontal scale from 0 to 10, with 0 indicating ''the worst score'' and 10 indicating ''the best score'', or with 0 indicating '''the best score'' and 10 indicating ''the worst score''.
Provider satisfaction | Through study completion, an average of 1 year
  Provider satisfaction, as measured by a self-developed Dutch provider satisfaction questionnaire, focuses on satisfaction about the intervention with the VR system or headphone with audio. The questionnaires included a Visual Analogue Scale (VAS). The VAS is a horizontal scale from 0 to 10, with 0 indicating ''the worst score'' and 10 indicating ''the best score'', or with 0 indicating '''the best score'' and 10 indicating ''the worst score''.
Change from baseline systolic blood pressure and diastolic blood pressure at 5 minutes after procedure | Baseline, 5 minutes after procedure
  The systolic blood pressure and diastolic blood pressure 5 minutes before the intervention (intervention group)/wound care (control group) and 5 minutes after the intervention (intervention group)/wound care (control group)
Change of systolic blood pressure and diastolic blood pressure during procedure | During procedure
  The systolic blood pressure and diastolic blood pressure every 5 minutes during procedure
Change from baseline blood oxygen level at 5 minutes after procedure | Baseline, 5 minutes after procedure
  The blood oxygen level, measured using a pulse oximetry device, 5 minutes before intervention (intervention group)/wound care (control group), and 5 minutes after the intervention (intervention group)/wound care (control group)
Change of blood oxygen level during procedure | During procedure
  The blood oxygen level every 5 minutes during procedure, measured using a pulse oximetry device
Change from baseline pulse rate at 5 minutes after procedure | Baseline, 5 minutes after procedure
  The pulse rate 5 minutes before intervention (intervention group)/wound care (control group), and 5 minutes after the intervention (intervention group)/wound care (control group)
Change of pulse rate during procedure | During procedure
  The pulse rate every 5 minutes during procedure
Change from baseline respiratory rate at 5 minutes after procedure | Baseline, 5 minutes after procedure
  The respiratory rate 5 minutes before intervention (intervention group)/wound care (control group), and 5 minutes after the intervention (intervention group)/wound care (control group)
Change of respiratory rate during procedure | During procedure
  The respiratory rate every 5 minutes during procedure

CONTACTS AND LOCATIONS:
Overall Officials: Marlies Schijven, Prof. dr., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam University Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No